CLINICAL TRIAL: NCT01516151
Title: A Randomized Open-label Dose-ranging, Multi-center Trial to Assess the Safety and Efficacy of NKPL66(CaPre™) in the Treatment of Mild-to-high Hypertriglyceridemia
Brief Title: Assess the Safety and Efficacy of NKPL66 (CaPre™) in the Treatment of Mild-to-high Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grace Therapeutics Inc. (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRT-API-NKPL66-CT-PIIB
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Hypertriglyceridemia
Keywords: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Active Comparator): 0.5g total CaPre™ from baseline to week 4 and 1.0g total CaPre™ from week 4 to week 8
  Interventions: Dietary Supplement: CaPre™
- Group B (Active Comparator): 1.0g total CaPre™ from baseline to week 4 and 2.0g total CaPre™ from week 4 to week
  Interventions: Dietary Supplement: CaPre™
- Group C (Active Comparator): 2.0g total CaPre™ from baseline to week 4 and 4.0g total CaPre™ from week 4 to week 8
  Interventions: Dietary Supplement: CaPre™
- Group D (Other): Standard of care
  Interventions: Drug: Lipid Lowering Medication
- Group E (Active Comparator): 4.0g total CaPre™ from baseline to week 8
  Interventions: Dietary Supplement: CaPre™

INTERVENTIONS:
Dietary Supplement: CaPre™ — 1 capsule of 0.5g total CaPre™ for 4 weeks followed by one 1.0g capsule per day for an additional 4 weeks
  Arms: Group A; Group B; Group C; Group E
Dietary Supplement: CaPre™ — 1 capsule of 1.0g total CaPre™ for 4 weeks followed by two 1.0g capsules per day for an additional 4 weeks
  Arms: Group A; Group B; Group C; Group E
Dietary Supplement: CaPre™ — 2 capsules of 1.0g total CaPre™ for 4 weeks followed by 4 capsules of 1.0g total per day for an additional 4 weeks.
  Arms: Group A; Group B; Group C; Group E
Drug: Lipid Lowering Medication — Patient will be treated as per the Standard of care.
  Arms: Group D
Dietary Supplement: CaPre™ — 4 capsules of 1 g total per day for 8 weeks.
  Arms: Group A; Group B; Group C; Group E

SUMMARY:
To evaluate the efficacy of 0.5, 1.0, 2.0 and 4.0 g/ day of CaPre™ in reducing fasting plasma serum triglycerides over a four week period in patients with mild-to-high hypertriglyceridemia as compared to the standard of care alone.

DETAILED DESCRIPTION:
The data generated from preclinical studies, as well as data accumulated from preclinical and clinical studies conducted with the precursor of CaPre™, NKO® , a natural health product (NPN: 80006416), have shown that CaPre™ is a safe product and well tolerated. In addition, there are preclinical data demonstrating that CaPre™ is effective in reducing circulating plasma concentrations of triglycerides. This effect is also accompanied by the regulation of other blood lipids, glucose tolerance and inflammatory biomarkers. These studies have been conducted in several preclinical adult phenotypes: (1) Healthy Sprague-Dawley (SD) rats, (2) obese and dyslipidemic Zucker Diabetic Fatty (ZDF) rats and(3-5) in three distinct murine phenotypes (normal wild-type C57BL/6, human ApoA-I transgenic mice and homozygous LDL-receptor knockout).

As the prevalence of cardiometabolic disorders progressively increase over the years, it is expected that there will be an augmentation in the necessity for new anti-dyslipidemic medications that can most importantly be added in combination to other treatments. Current treatment methods address a specific target indication, but do not offer complete management of dyslipidemia.

We are now left with the option to either inadequately treat patients suffering from cardiovascular and metabolic disorders or, to prescribe combination treatments hoping to address the risk factors while mitigating their known side effects. A treatment gap exists since there is no medication that increases HDL-cholesterol and reduces triglycerides while reducing LDL-cholesterol without side effects.

At present there is a need to assess the effectiveness of CaPre™ in reducing triglycerides in patients with high hypertriglyceridemia. The current study will address these issues and will generate the evidence that will be required to determine whether this product could be effectively used in the clinical management of this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18 to 75 years;
* Fasting plasma levels of TG > 2.28 and < 10 mmol/L (200 and 877 mg/dL) on two occasions within 2 weeks (screening and baseline/part 1 visits).
* Patients who are currently not on pharmacotherapy for hyperlipidemia and according to the judgement of the physician and Canadian Guidelines for the Diagnosis and Treatment of Dyslipidemia initiation of drug therapy is not indicated for the duration of the study.

OR

* Patients currently treated with statins and according to the judgement of the physician and the Canadian Guidelines for the Diagnosis and Treatment of Dyslipidemia a change in their current drug regimen is not indicated for the duration of the study.
* Patients treated with statin must be on stable dose for at least 6 weeks prior to screening;
* Patients are willing to follow the NCEP Step 1 Diet (see Appendix 4) for the duration of the study;
* Female participants of childbearing potential (i.e. not surgically sterilized or post-menopausal greater than one year) must have negative serum pregnancy test and must be using an effective birth control method, defined as:

  * continuous use of oral or long acting injected contraceptive for at least 2 months prior to study entry, or;
  * use of an intra-uterine device or implantable contraceptive, or;
  * use of double barrier methods of birth control

Exclusion Criteria:

* Any concomitant medication which in the opinion of the investigator would preclude the patient from successfully participating in the study;
* Women who are pregnant or that are breast feeding;
* Participation in another clinical trial within 30 days from initiation of the study;
* Participants with a high risk for cardiovascular disease; (The definition of high-risk individuals will follow that of the 2009 Canadian Guidelines and include a) FRS >= 20% 10-year risk; b) All patients with uncontrolled diabetes (DCA guidelines) and c) Evidence of atherosclerosis -when this evidence was ascertained when clinically indicated);
* Systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg. In diabetic patients, systolic blood pressure > 130 mmHg and/or diastolic blood pressure > 90 mmHg.
* History of stroke, intermittent claudication or transient ischemic attack;
* Known unstable (uncontrolled) cardiac disease, within the last 6 months:
* Patient with a clinically significant abnormal ECG at screening.
* Patients with uncontrolled diabetes mellitus, with HbA1c > 7.0%;
* Known diagnosis of hypoglycemia
* Evidence of active renal disease indicated by a fasting estimated glomerular filtration rate (eGFR) of < 60 ml/min per 1.73 m2;
* Increased plasma levels (>ULN) of amylase (as per respective lab upper limits) and / or lipase (>160 IU/L) or any indication of pancreatitis (increased alcohol consumption, gallstones);
* History of pancreatitis;
* Use of any lipid lowering medication other than statins (e.g niacin, fibrates or ezetimibe) and/or lipid lowering NHP within 6 weeks prior to the screening visit;
* Intake of > 2 servings per week of fish or regimented use of fish oil/omega-3 supplements within 6 weeks prior to the screening visit;
* Intake of fortified foods containing plant sterols within 6 weeks prior to the screening visit;
* Known HIV or Hepatitis B or C positive;
* Patients with osteoporosis and hormone sensitive conditions;
* Patients with uncontrolled asthma as defined by the 2010 Consensus Summary of the Canadian Thoracic Society;
* Known seafood allergy or allergy to any of the medicinal or non-medicinal ingredients of the study medication, including:

  * Omega-3 fatty acids (including EPA and DHA)
  * Phospholipids (mainly phosphatidylcholine)
  * Astaxanthin
  * Bovine gelatin
* Coagulopathy or on anticoagulants. Platelet aggregation inhibitors (such as aspirin or clopidogrel but not heparin) are permitted in the study; patients taking both aspirin and clopidogrel are not permitted in the study;
* Unable or unwilling to comply with the protocol;
* Patient reported weight must be stable for the past 6 months (within 3kg variation);
* Consumption of more than 14 standard alcoholic drinks a week.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Percent change in fasting blood circulating serum TGs | Between baseline and 4 weeks of treatment.
  The percent change in fasting blood circulating serum TGs between baseline and 4 weeks of treatment.

SECONDARY OUTCOMES:
Absolute change in fasting plasma TGs | Baseline, Week 4 and Week 8
  Absolute change in fasting plasma TGs;
Patients achieving target TG fasting plasma levels | Baseline
  Percentage (%) of patients achieving target TG fasting plasma levels (TG<1.7 mmol/L);
Change in fasting plasma LDL-C, VLDL-C, HDL-C, total cholesterol, hs-CRP and non-HDL | Between baseline and 4 and 8 weeks of treatment
  Absolute change in fasting plasma LDL-C, VLDL-C, HDL-C, total cholesterol, hs-CRP and non-HDL
Change in fasting plasma concentrations of LDL-C, VLDL-C, HDL-C, total cholesterol, hs-CRP and non-HDL | Between baseline and 4 and 8 weeks of treatment
  Percentage (%) change in fasting plasma concentrations of LDL-C, VLDL-C, HDL-C, total cholesterol, hs-CRP and non-HDL;
Calculated ratios | The percent change in fasting blood circulating serum TGs Between baseline and 4 and 8 weeks of treatment.
  Calculated Ratios:
  1. Total cholesterol : HDL-C
  2. LDL-C : HDL-C
  3. TGs : HDL-C
Change in fasting plasma concentrations of biomarkers | Between baseline and 4 and 8 weeks of treatment
  Absolute and percent (%) change in fasting plasma concentrations of biomarkers;
  1. Glycated Hemoglobin (HbA1c)
  2. Glucose
  3. Creatinine phosphokinase (CPK)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dufour, M.D., Principal Investigator — Institut de Recherches Cliniques de Montreal
Locations (38):
- Canada (38):
  - Alberta Health Services Clinical Trials, Red Deer, Alberta
  - Abbotsford, British Columbia
  - Kelowna, British Columbia
  - BC Diabetes, Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Dieppe, New Brunswick
  - Entralogix Clinical Research, Aurora, Ontario
  - Entralogix Clinical Research, Brampton, Ontario
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - Thamesview Ctr of Family Med, Chatam, Ontario
  - Moran Medical Centre, Colingwood, Ontario
  - C & L Research, Fort Erie, Ontario
  - G.S. Cardiac Lab Medicine Professional Corp, Greater Sudbury, Ontario
  - Hamilton, Ontario
  - Entralogix Clinical Research, Kitchener, Ontario
  - Entralogix Clinical Research, Mississauga, Ontario
  - Malton Medical Research Group, Mississauga, Ontario
  - Niagara Falls, Ontario
  - Entralogix Clinical Research, North York, Ontario
  - Taunton Health Centre, Oshawa, Ontario
  - Steeple Hill Medical centre, Pickering, Ontario
  - Entralogix Clinical Research, Toronto, Ontario
  - Eric Silver Medicine Professional Corporation, Toronto, Ontario
  - Clinique Médicale des Trois Lacs, Vaudreuil Dorion, Ontario
  - Clinique Medicale Valcartier, Courcelette, Quebec
  - Clinique Reseau le Trait d'Union, Delson, Quebec
  - Clinique Medicale Mistassini, Dolbeau-Mistassini, Quebec
  - Clinique medicale, Grand-Mère, Quebec
  - GMF Grand Mere, Grand-Mère, Quebec
  - CRM Lanaudiere, Joliette, Quebec
  - Applied Medical Information Research AMIR, Montreal, Quebec
  - Centre de recherche A&E, Québec, Quebec
  - Clinique des maladies lipidiques de Quebec Inc., Québec, Quebec
  - Clinique Services Sante Rosemere, Rosemère, Quebec
  - Csss de St-Jerome, Saint-Jérôme, Quebec
  - CSSS Vallee De L'Or, Val-d'Or, Quebec
  - Applied Medical Information Research (AMIR), Westmount, Quebec

REFERENCES:
- [Derived] Kim KS, Belley-Cote EP, Walsh M, Wang A, Balasubramanian K, Treleaven N, Garg AX, Guyatt G, Whitlock RP. Left atrial appendage occlusion study III-Kidney substudy. Am Heart J. 2025 Oct;288:90-100. doi: 10.1016/j.ahj.2025.04.018. Epub 2025 Apr 19. PMID 40258408